CLINICAL TRIAL: NCT05841810
Title: Scaling and Sustaining COVID-19 Vaccination Through Meaningful Community Engagement and Care Coordination for Underserved Communities
Brief Title: Working Towards Empowered Community-driven Approaches to Increase Vaccination and Preventive Care Engagement
Acronym: WEAVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Ysidro Health Center (Other)
Responsible Party: Principal Investigator, Nicole Stadnick, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01MD017222 (NIH)
Record Dates: First submitted 2023-03-28; First posted 2023-05-03 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: COVID-19
Keywords: implementation science; hybrid 3 effectiveness-implementation study; sequential multiple assignment randomized trial; COVID-19; underserved communities; health equity; care coordination; mHealth; preventive care
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The investigators will use a hybrid type 3 effectiveness-implementation sequential multiple assignment randomized trial (SMART) design to assess the impact of our multicomponent health program on implementation and outcome measures. As participants progress through multiple stages, each participant may be randomized to two or more intervention options allowing us to compare the relative effectiveness of multiple intervention options. Our experimental design follows a SMART randomized structure to introduce the more intensive care coordination component only to those who are not responding to usual care or the lower intensity and less resource intensive mHealth messaging component allowing for more efficient resource allocation.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Stage 1 mHealth Outreach (Experimental)
  Interventions: Other: mHealth Outreach
- Stage 2 mHealth Outreach (Experimental)
  Interventions: Other: mHealth Outreach
- Stage 1 Standard of Care (No Intervention)
- Stage 2 Standard of Care (No Intervention)
- Stage 2 mHealth Outreach + Care Coordination (Experimental)
  Interventions: Other: mHealth Outreach; Other: Care Coordination

INTERVENTIONS:
Other: mHealth Outreach — Community outreach using mHealth messaging will be led by community weavers via SMS and voice messages about COVID-19 vaccines and preventive care engagement in languages spoken by patients (i.e., Spanish, Arabic, Vietnamese).
  Arms: Stage 1 mHealth Outreach; Stage 2 mHealth Outreach; Stage 2 mHealth Outreach + Care Coordination
Other: Care Coordination — Inclusive of standard of care coordination with added focus on completing outstanding preventive care practices. Care coordination will be focused on collaborative problem-solving and case management to help patients schedule and attend recommended annual preventive health care, including a routine physical exam, recommended preventive screenings and COVID-19 vaccination
  Arms: Stage 2 mHealth Outreach + Care Coordination

SUMMARY:
This study will optimize, implement, and test the impact of our multicomponent health program that includes three primary implementation strategies (Cultural Weavers and co-creation, mHealth strategies using culturally meaningful text and voice messages, and care coordination). The investigators will use a participatory approach to engage community members in co-creating and optimizing our mHealth outreach and enhanced care coordination program components. The investigators will use a hybrid type 3 effectiveness-implementation sequential multiple assignment randomized trial (SMART) design to assess the impact of our multicomponent health program on implementation and outcome measures.

DETAILED DESCRIPTION:
This is an adaptive intervention which utilizes a multi-component messaging and care coordination to increase COVID19 vaccine uptake.

Aim 1: Optimize a multicomponent health program to promote COVID-19 vaccine uptake and engagement in preventive healthcare using our established co-creation approach to address multi-level (individual, community, systemic) barriers to vaccine uptake and preventive care engagement.

Community engagement through Community Advisory Boards and Community Weavers. The multicomponent health program will be developed and optimized using our established co-creation approach with guidance from Community Weavers and engagement of the community through Community Advisory Boards (CABs). Hiring criteria for Community Weavers will include that they are fluent in at least one of the three priority languages (i.e., Spanish, Arabic, Vietnamese) and have at least six months of community organizing, leading, or community engagement experience. Community Weavers will have a critical role in developing and refining the tailored mHealth messages. They will also be instrumental in facilitating the existing care coordination efforts at the FQHC by focusing on immigrant and refugee communities that can be difficult to engage in care. The Community Weavers will also lead three CABs that each include five members inclusive of the three primary languages spoken by community members of our clinics of interest will be invited to participate.

During the first year, each CAB will meet monthly or twice monthly up to four times (two hours per meeting). These initial CAB meetings will be charged with co-creating content and frequency for the mHealth outreach (SMS and voice messages) and identifying topics to be covered in and strategies and processes for the care coordination program. To facilitate mHealth message development, Cultural Weavers will use a story telling/narrative framework approach inviting residents to join open dialogue and share their journey through the decision-making process towards getting vaccinated, reflecting on the anxieties they navigated, the misinformation they were confronted with, and any structural or technological barriers they had to overcome to enhance the cultural resonance and tailoring of the mHealth messages.90 In subsequent years, the CABs will continue meeting quarterly to revise and update mHealth content and engage in an Appreciative Inquiry Process to evaluate the implementation of the multicomponent health program and determine when refinements for optimization are needed to both the mHealth and care coordination components. The co-creation and optimization of the program components will be guided by the contextual domains of PRISM (i.e., Intervention characteristics, Recipient characteristics, Implementation and sustainability infrastructure, External environment) and will build on our prior work with the community and the CAB members' lived experience as members of the respective communities.

Throughout the project, the investigators will evaluate the quality and extent of stakeholder engagement using a concurrent (QUAN + QUAL) mixed methods approach that the investigators developed through our NIH funded COVID-19 projects. The investigators will implement a stakeholder engagement survey completed via online distribution by all stakeholders following each CAB meeting using the Goodman et al. 9-item measure inquiring about how well and how frequently eight engagement principles were perceived during the meeting and an open-ended reflection question. Ethnographic documentations of the CAB process will be conducted by trained research staff and will use our structured documentation form that identifies various aspects of engagement (e.g., topics covered, interruptions, time spent contributing). Survey data will be summarized as simple frequencies and text responses will be coded using an open coding approach. Data from the documentation rubrics will be abstracted using a matrix approach the investigators developed in our prior work and will be triangulated with information from the survey. Survey information will be reviewed after each CAB meeting and used to support the iterative improvement of the CAB processes.

mHealth Outreach. Specific mHealth messaging will include personalized SMS and automated phone calls recorded by community leaders in their respective languages aligned with the language preferences of our target SYH clinics. The content of the mHealth outreach will include information about how and where to get COVID-19 vaccinated, COVID-19 vaccine side effects, the importance of and timing of priority preventive services, and how to schedule those services, as well as dispelling myths about vaccines and providing reminders for appointments. mHealth content and distribution frequency will be determined by each Community Advisory Board to align with their community's preferences and needs. It is expected that 1-2 voice and/or SMS messages will be delivered weekly to the Aim 2 sample. New messages will be developed and added to our message library based on updated public health guidance and feedback from our participants. Our mHealth outreach system will be user tested and refined prior to Aim 2 launch.

Care Coordination. Care coordination will be focused on collaborative problem-solving and case management to help patients schedule and attend recommended annual preventive health care, including a routine physical exam, recommended preventive screenings (e.g., mammograms, A1c screening, colorectal cancer screening), and COVID-19 vaccination. SYH has an established process to provide care coordination and the investigators will refine these processes (e.g., eligibility, health education topics, duration of care coordination) through input from our Community Advisory Board. For this study, SYH will hire study-specific care coordinators who are members of the three communities represented by the Community Advisory Board. Care coordination will be tailored to the needs and cultural preferences of the respective patient community. The content of care coordination will include initial engagement and re-engagement of patients in preventive care services, developing a patient health action plan, support with adhering to the health action plan, scheduling preventive care appointments, and communicating with the patient's care team to ensure continuity of care.

Aim 2: Evaluate the implementation, effectiveness, and sustainment of the multicomponent COVID-19 vaccine and preventive care engagement program using a hybrid type 3 implementation-effectiveness sequential multiple assignment randomized trial design across immigrant, refugee, Latino, and BIPOC communities in Central and East San Diego.

A total of 300 patients (100 per clinic), from a sampling frame of approximately 5000 patients, will be recruited to participate in the study. Recruitment will be from all language groups, and the investigators will work with CABs to develop culturally appropriate recruitment methods to ensure participation from all three language groups (i.e., Spanish, Arabic, and Vietnamese). The investigators will consider a weighted sampling approach if patient volume varies considerably between the three clinics during the baseline period. While these language groups are broad, they are all connected with the partnering FQHC, which helps frame the target populations for this research project. Furthermore, to understand reach for our program, the investigators will document the characteristics of those participating in the study and compare it to the population in each of the three geographic regions recruited into the study (Community Heights, El Cajon, Escondido).

Patient recruitment will occur at each of the three participating SYH clinics through collaborative efforts between the SYH Care Coordinators, Global ARC Cultural Weavers, and UC San Diego Health and Technology Specialists. This is an adaptive intervention which utilizes a multi-component messaging and care coordination to increase COVID19 vaccine uptake. Both randomization and analysis will be conducted at the individual participant level. The hybrid type 3 trial will span 4 years inclusive of two years of active implementation and 2 years of sustainment/maintenance. At enrollment, participants will be stratified by current COVID-19 vaccination status, then randomized into the first stage intervention (mHealth outreach or standard of care). Response or lack of response after the completion of the first stage intervention will determine if participants continue in their initial first stage intervention or re-randomized to increased intensity intervention. Non-responders in the standard of care arm will be equally re-randomized into either mHealth outreach or enhanced care coordination for stage 2. Non-responders in mHealth outreach will be re-randomized into mHealth or mHealth plus enhanced care coordination for stage 2. Non-response will be defined as not being up to date on COVID-19 vaccination OR having at least one outstanding preventive care need.

Data collection and measures. Data will be collected using multiple sources to represent diverse perspectives using a QUANT+QUAL concurrent (mixed method design approach). Data sources include data from delivery of the core components of the program, data from participants, and EHR clinical outcomes data. Surveys and interviews with participants will be conducted in the participant's preferred language. Interviews will be led by Community Weavers. Study databases for mHealth message delivery, care coordination, and Community Weavers will be in REDCap surveys allowing for the entry of real time information. Periodic reflections will be collected as weekly diary entries from different members of the research team and notes from monthly meetings reviewing these entries. Participant surveys will be drafted with input from the CABs and pilot tested prior to full implementation. A combination of electronic and paper-based surveys based on the preference of the participants will be used.. Interviews will be conducted by the Community Weavers using a semi-structured interview guide reflecting PRISM domains adapted from prior studies and vetted by the CAB.

This 5-year R01 NIMHD proposal capitalizes on the unique and complementary methods from community engagement, implementation science, health equity, health communication, infectious disease, and public health to co-create a multicomponent health program to promote sustained COVID-19 vaccination and preventive care engagement for underserved communities in San Diego. This proposal extends current work using a generalizable co-creation approach and funded by NIH CEAL and RADx-UP initiatives to focus on scaling and sustaining COVID-19 and broader health equity for immigrant, refugee, and BIPOC communities. Limited research exists on sustainment strategies so the explicit focus on scaling and sustaining will add to the field of implementation science by adding evidence to health equity-promoting sustainment strategies. Results from this study will be used to develop a multi-site scaling out study in a subsequent NIH R01 application.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Speaks Spanish, Arabic and/or Vietnamese.
* Current San Ysidro Health patient and receives care at select clinics in study locations (Escondido, El Cajon, Community Heights).

Exclusion Criteria:

* Not able to provide informed consent.
* < 18 years old
* Does not speak Spanish, Arabic or Vietnamese
* Is not a current San Ysidro Health patient or is a current San Ysidro Health patient but does not receive care at select clinics in study locations (Escondido, El Cajon, Community Heights).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccination rate | 8 months after starting the 1st stage intervention to determine response vs non-response for 2nd stage randomization.
  Clinical assessment of COVID-19 vaccine status based on the total number of COVID-19 vaccines received (initial + boosters).
COVID-19 vaccination rate | 12 months after 2nd stage randomization
  Clinical assessment of COVID-19 vaccine status based on the total number of COVID-19 vaccines received (initial + boosters).
COVID-19 vaccination rate | 24 months after 2nd stage randomization
  Clinical assessment of COVID-19 vaccine status based on the total number of COVID-19 vaccines received (initial + boosters).
COVID-19 vaccination rate | 36 months after 2nd stage randomization
  Clinical assessment of COVID-19 vaccine status based on the total number of COVID-19 vaccines received (initial + boosters).

SECONDARY OUTCOMES:
Preventive services engagement rate | 8 months after starting the 1st stage intervention to determine response vs non-response for 2nd stage randomization.
  Secondary effectiveness outcomes will be an increase in preventive service engagement defined as completing a physical exam and at least one recommended preventive care screening (e.g., mammogram, A1c screening, colorectal cancer screening, blood pressure screenings).
Preventive services engagement rate | 12 months after 2nd stage randomization
  Secondary effectiveness outcomes will be an increase in preventive service engagement defined as completing a physical exam and at least one recommended preventive care screening (e.g., mammogram, A1c screening, colorectal cancer screening, blood pressure screenings).
Preventive services engagement rate | 24 months after 2nd stage randomization
  Secondary effectiveness outcomes will be an increase in preventive service engagement defined as completing a physical exam and at least one recommended preventive care screening (e.g., mammogram, A1c screening, colorectal cancer screening, blood pressure screenings .
Preventive services engagement rate | 36 months after 2nd stage randomization
  Secondary effectiveness outcomes will be an increase in preventive service engagement defined as completing a physical exam and at least one recommended preventive care screening (e.g., mammogram, A1c screening, colorectal cancer screening, blood pressure screenings).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - San Ysidro Health Medical Center - El Cajon, El Cajon, California
  - Escondido Family Medicine, Escondido, California
  - University of California San Diego, La Jolla, California
  - Community Heights Family Medicine, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stadnick NA, Geremia C, Cain KL, Oswald W, Watson P, Ibarra M, Nguyen M, Altemimi Z, Hammi N, Bautista M, Alrefaee M, Chu TM, Wagner NM, Vijaykumar S, O'Leary ST, Diaz EA, Aldous J, Rabin BA. Illustrating Key Components to Co-Creation Through Preventive Care mHealth Messaging with Underserved Communities and Expert Partners. J Med Syst. 2025 Dec 12;49(1):180. doi: 10.1007/s10916-025-02310-z. PMID 41381776
- [Derived] Rabin BA, Cain KL, Watson P Jr, Oswald W, Laurent LC, Meadows AR, Seifert M, Munoz FA, Salgin L, Aldous J, Diaz EA, Villodas M, Vijaykumar S, O'Leary ST, Stadnick NA. Scaling and sustaining COVID-19 vaccination through meaningful community engagement and care coordination for underserved communities: hybrid type 3 effectiveness-implementation sequential multiple assignment randomized trial. Implement Sci. 2023 Jul 14;18(1):28. doi: 10.1186/s13012-023-01283-2. PMID 37443044